CLINICAL TRIAL: NCT07068347
Title: Comparison Of Virtual Reality And Conventional Physical Therapy, With And Without Life Style Modification, On Upper Limb Dysfunction In Post-Surgical Breast Cancer Survivors
Brief Title: Comparison Of VR & CPT, With And Without Lifestyle Modification, On ULD In Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PhDRSW/Batch-Fall23/2223
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Lottery method into four groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR + lifestyle modification (Experimental)
  Interventions: Combination Product: VR + lifestyle modification
- VR only (Active Comparator)
  Interventions: Combination Product: VR only
- Conventional physical therapy + lifestyle modification (Active Comparator)
  Interventions: Combination Product: Conventional physical therapy + lifestyle modification
- Conventional physical therapy only (Active Comparator)
  Interventions: Combination Product: Conventional physical therapy only

INTERVENTIONS:
Combination Product: VR + lifestyle modification — VR + lifestyle modification (Warm up,In VR kinetic sports I Bowling, Darts,Golf,Boxing,Beach Volleyball ,Table Tennis,Fruit Ninja)Passive glenohumeral joint mobilization,Scar tissue massage.In lifestyle modification walking at home for 30 min in 3-5 days /week. Dietry habits will be given according to American Institute for cancer Research.
  In sleep habits Recommended Sleep Hours 7-9 hours per night,Establish a Consistent Sleep Schedule,Create a Comfortable Sleep Environment,Limit Screen Time Before Bed,Engage in Relaxation Techniques,Limit Caffeine and Alcohol Intake,Manage Nighttime Discomfort,Maintain a Pre-Sleep Routine,Address Emotional Health,Avoid Daytime Naps.Deep breathing exercise for stress management
  Arms: VR + lifestyle modification
Combination Product: VR only — VR only (Warm up,In VR kinetic sports I Bowling, Darts,Golf,Boxing,Beach Volleyball ,Table Tennis,Fruit Ninja)Passive glenohumeral joint mobilization,Scar tissue massage.
  Arms: VR only
Combination Product: Conventional physical therapy + lifestyle modification — Conventional physical therapy + lifestyle modification In Conventional physical therapy(Pumping exercise for upper limb,Pendulum exercises ,Shrugs for shoulder and rotations,In sitting position arms up with clasped hands ,Shoulder rotation (arms on sides-arms in abduction),Arms up with hands clasped again but in lying position ,Wand exercises ,M. pectoralis major-M. Pectoralis Minor stretches in supine and standing positions,Snow angels,Front and lateral climbing on wall ,Trunk rotation in standing position (in sitting position, if not tolerated)
  Arms: Conventional physical therapy + lifestyle modification
Combination Product: Conventional physical therapy only — Conventional physical therapy only((Pumping exercise for upper limb,Pendulum exercises ,Shrugs for shoulder and rotations,In sitting position arms up with clasped hands ,Shoulder rotation (arms on sides-arms in abduction),Arms up with hands clasped again but in lying position ,Wand exercises ,M. pectoralis major-M. Pectoralis Minor stretches in supine and standing positions,Snow angels,Front and lateral climbing on wall ,Trunk rotation in standing position (in sitting position, if not tolerated) ,Trunk lateral flexion with arms in 90 degrees abduction in standing position,Theraband (flexion-extension-abduction, adduction and internal-external rotation),Muscles of upper limb strengthening ,Mobilization for passive glenohumeral joint ,Tissue massage for scars.
  Arms: Conventional physical therapy only

SUMMARY:
The proposed study will compare the effect of an application of non-immersive virtual reality (VR) and conventional physical therapy (CPT) with and without lifestyle changes on upper limb dysfunction in breast cancer survivors, post-surgery. The purpose of this proposed RCT is to compare the effect of VR alone/in conjunction with lifestyle changes to that of CPT alone/in conjunction with lifestyle changes for the physical rehabilitation of female breast cancer survivors. Research will be conducted on 60 patients. This research employs parallel, randomized clinical trial design, which shall be conducted in NORI hospital, Shifa International Hospital and Kinifit physiotherapy in Islamabad/Rawalpindi over a period of 18 months. Thus, the type of sampling done in this study is purposive sampling.

DETAILED DESCRIPTION:
Primary Objectives:

1. To compare the effects of immersive virtual reality and conventional physical therapy, with and without lifestyle modification, on upper limb functional disability in post-surgical breast cancer survivors.

   Secondary Objectives:
2. To assess the effects of immersive virtual reality compared to conventional physical therapy, with and without lifestyle modification, on improving pain, shoulder range of motion and muscle strength in post-surgical breast cancer survivors.
3. To determine the effects of immersive virtual reality compared to conventional physical therapy with and without lifestyle modification on quality of life and psychological wellbeing in post-surgical breast cancer survivors.
4. To evaluate self-reported adherence to the life style modification program among post-surgical breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivors aged 30-60 years.
* Women with breast cancer who have undergone any type of breast cancer surgery (e.g., mastectomy, lumpectomy, or breast reconstruction), regardless of the specific surgical procedure will be included.
* Participants able to carry on upper limb and whole-body physical activity will be included.
* Participants able to use smart devices such as mobile phones and computers will be included.
* Patients obtaining a physician's clearance for fitness testing and exercise will be included.
* Patients having no physical limitations prohibiting exercise will be included.
* Patients diagnosed with grade 0-3 of breast cancer who had undergone surgery will be included.
* who were currently in the 2nd ~ 4th months after cancer surgery.
* Presence of upper limb dysfunction (e.g., pain, reduced range of motion and weakness).

Exclusion Criteria:

* Subjects suffering from active malignant tumors or bilateral breast cancer.
* Participants disabling physical or psychological ailments not allowing them to participate in the intervention .
* Patients who had lymphedema will be excluded.
* Participants with visual disorders that interfered with a video game- based exercise.
* Subjects with cognitive disorders, mental disorders, or cooperation issues will be excluded.Subjects with vascular or cardiopulmonary disorders.
* Subjects with previous breast cancer surgery on the present or contralateral side.
* Participants having upper extremity ROM limitation before the surgery will be excluded.
* Participants with presence of pace-maker, infection, open wounds, or wound drains will be excluded.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 18 Months
  Upper limb dysfunction can be assessed using a combination of pain evaluation, range of motion measurements, and muscle strength testing. Pain is typically recorded using the Visual Analog Scale (VAS), where the patient marks their perceived pain level along a 10-centimeter horizontal line, with 0 indicating no pain and 10 representing the worst imaginable pain.
Goniometer (shoulder flexion, abduction, external rotation) | 18 Months
  Scoring details: The score is determined by measuring the distance in centimeters from the 'no pain' end to the patient's mark. Range of motion (ROM) is assessed using a goniometer for key movements such as shoulder flexion, abduction, and external rotation. The angles achieved are measured in degrees and compared against established normative values typically 0° to 180° for flexion and abduction, and 0° to 90° for external rotation to identify limitations.
Handheld dynamometer | 18 Months
  Muscle strength is evaluated using a handheld dynamometer, measuring the force produced by muscle groups like shoulder flexors, abductors, and external rotators. Strength is recorded in kilograms or newtons, usually averaging three trials, and compared to normative data or the unaffected limb to determine the degree of weakness. Together, these measures provide a comprehensive functional profile of the upper limb.
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | 18 Months
  Functional outcomes for individuals with upper limb dysfunction can be evaluated using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, a widely used, standardized, self-reported measure. The DASH consists of 30 items that assess the patient's ability to perform various physical activities, severity of symptoms, and impact on social and work-related tasks involving the upper extremity. Each item is rated on a 5-point Likert scale, ranging from 1 (no difficulty or no symptoms) to 5 (unable to perform activity or extreme symptoms). The scores from all completed items are summed, averaged, and then transformed into a score out of 100, where 0 indicates no disability and 100 represents the most severe disability. This tool provides valuable insight into the patient's perceived functional status and the extent to which upper limb issues interfere with daily life and occupational tasks.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 18 Months
  his is a validated, multidimensional, self-administered questionnaire designed to evaluate overall health-related quality of life in patients with chronic illness or undergoing treatment. The QLQ-C30 consists of 30 items covering several domains, including five functional scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), a global health status/quality of life scale, and several single-item assessments for additional symptoms such as insomnia, appetite loss, and financial difficulties. Each item is rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much), except for the two global health status items, which use a 7-point scale. Scores are transformed to a scale from 0 to 100, with higher scores on the functional and global health scales indicating better functioning and quality of life, while higher scores on the symptom scales reflect greater symptom burden.
Hospital Anxiety and Depression Scale (HADS) | 18 Months
  The HADS consists of 14 items, divided equally into two subscales: seven items assess symptoms of anxiety (HADS-A) and seven assess symptoms of depression (HADS-D). Each item is scored on a 4-point Likert scale ranging from 0 to 3, with total scores for each subscale ranging from 0 to 21. Scores are interpreted as follows: 0-7 indicates a normal range, 8-10 suggests possible anxiety or depression, and 11-21 indicates probable or clinically significant anxiety or depression.
Self-reported adherence to the lifestyle modification program through weekly logs. | 18 Months
  The Health-Promoting Lifestyle Profile II (HPLP-II) is scored using a 4-point Likert scale (Never, Sometimes, Often, Routinely) for each of its 52 items. The overall score is calculated as the mean of all item responses, and this mean score is then categorized into four levels: Poor, Moderate, Good, and Excellent. The collected data provides insight into patient engagement, consistency in following health recommendations, and potential barriers to adherence. Regular review of these weekly logs allows clinicians or researchers to track progress, identify patterns of non-compliance, and offer timely support or program adjustments to improve health behaviors and functional recovery outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - District Head Quarters Hospital, Rawalpindi, Punjab Province
  - Holy Family Hospital, Rawalpindi, Punjab Province
  - Kinifit Physiotherapy Center, Islamabad

IPD SHARING:
Plan to Share IPD: No